CLINICAL TRIAL: NCT05253170
Title: A Randomized Phase III Trial of Hypofractionated Versus Conventionally Fractionated Radiotherapy in Breast Cancer Patients With Reconstruction After Mastectomy
Brief Title: Hypo Versus Conventional Fractionation in Reconstructed-Breast Cancer Mastectomy Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, In Ah Kim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KROG 21-07
Record Dates: First submitted 2022-02-15; First posted 2022-02-23 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer; Radiotherapy; Complications
Keywords: Mastectomy; Reconstruction; Radiation therapy; Conventional fractionation; Hypofractionation; Complication
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionation (Experimental): For the cumulative total dose of 39-45.9 Gy to the chest wall, a daily dose of 2.5-3.0 Gy is administered 13-17 fractions.
  * Should be started within 3 months of completion of mastectomy or chemotherapy.
  * Clinical target volume (CTV) may include regional lymph nodes.
  * If a tissue expander or implant is present at the time of radiotherapy planning, CTV contouring should be performed according to the ESTRO ACROP implant-based target delineation guidelines.
  Interventions: Radiation: Hypofractionation
- Conventional Fractionation (Active Comparator): For the cumulative total dose of 45-50.4 Gy to the chest wall, a daily dose of 1.8-2.0 Gy is administered 23-28 fractions.
  * Should be started within 3 months of completion of mastectomy or chemotherapy.
  * Clinical target volume (CTV) may include regional lymph nodes.
  * If a tissue expander or implant is present at the time of radiotherapy planning, CTV contouring should be performed according to the ESTRO ACROP implant-based target delineation guidelines.
  Interventions: Radiation: Conventional Fractionation

INTERVENTIONS:
Radiation: Hypofractionation — Radiation regimen of 2.5-3.0Gy x 13-17 fractions +/- sequential boost 0-7 fractions
  Arms: Hypofractionation
Radiation: Conventional Fractionation — Radiation regimen of 1.8-2.0Gy x 23-28 fractions +/- sequential boost 0-5 fractions
  Arms: Conventional Fractionation

SUMMARY:
This randomized Phase III study aims to show major complication rate of hypofractionation radiation therapy is not inferior, compared to conventional fractionation radiation therapy in breast cancer patients undergoing mastectomy and reconstruction surgery.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, phase 3 clinical trial. For breast cancer patients who underwent breast reconstruction after mastectomy, the hypofractionation radiotherapy group (experimental group) and the conventional fractionation radiotherapy group (control group) were divided 1:1 and compared to reveal the non-inferiority with hypofractionation in terms of major complication rate.

I. Primary Objective

* To show the non-inferiority of major complication rate in reconstructed-breast between the hypofractionation radiotherapy group (experimental group) and the conventional fractionation radiotherapy group (control group) at 2 years after radiation therapy.
* The main complications are defined at those requiring hospitalization or surgery among complications.

II. Secondary Objective:

* Comparison of other side effects between the two groups.
* Comparison of complication rate stratified by reconstruction timing and type of reconstruction

  * Immediate implant-based reconstruction
  * Immediate autologous reconstruction
  * Delayed-immediate implant reconstruction (2-stage)
* Comparison of quality of life between the two groups.
* Comparison of local and regional control rates between the two groups.

III. Tertiary Objective:

* Comparison of cosmetic evaluations between the two groups.
* Dosimetry analysis for correlation between the occurrence of complications and the dose profile.

ELIGIBILITY:
Inclusion Criteria:

* Female patient who underwent mastectomy for invasive breast cancer
* Patients who have undergone breast reconstruction after mastectomy or who have inserted a tissue expander
* (y)p patients with stage IIIA or lower (excluding T4 and N3 patients) who need adjuvant radiation therapy
* Eastern Cooperative Oncology Group Performance ≤ 2
* Age ≥ 19 years
* Patients who agreed to participate in the study

Exclusion Criteria:

* Patients who already had implants at the time of diagnosis of breast cancer or who have already undergone reconstructive surgery
* Patients who underwent reconstruction after partial resection or breast conserving surgery rather than mastectomy
* Patients who are using or planning to use an air expander
* Patients receiving radiation therapy for salvage or palliative purposes
* Patients with distant metastases at the time of diagnosis
* Patients who are scheduled to undergo concurrent chemoradiation therapy
* Patients with bilateral breast cancer
* Male breast cancer patients
* Patients who have previously received radiation therapy for the ipsilateral breast or supraclavicular area
* Patients with history of cancers other than thyroid cancer, intraepithelial cancer of the cervix, or skin cancer
* Patients diagnosed with ductal breast carcinoma in situ, lobular carcinoma in situ, phyllodes, metaplastic cancer, or other benign tumors based on histological diagnosis

Ages: 19 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 622 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Complication Rate | Up to 2 years after the completion of radiation therapy
  * Unplanned re-hospitalization or re-operation for intervention
  * Implant removal due to infection, autologous flap total failure (reconstruction failure)
Capsular Contracture (If implant-based recontruction is performed) | Up to 2 years after the completion of radiation therapy
  • Baker Scale
  * G1: the breast is normally soft and appears natural in size and shape
  * G2: the breast is a little firm, but appears normal
  * G3: the breast is firm and appears abnormal
  * G4: the breast is hard, painful to the touch, and appears abnormal

SECONDARY OUTCOMES:
Hematoma | Up to 2 years after the completion of radiation therapy
  NIH-NCI Common Terminology Criteria for Adverse Events (CTCAE) Ver.5.0
  * G1: Mild symptoms; intervention not indicated
  * G2: Minimally invasive evacuation or aspiration indicated
  * G3: Transfusion; invasive intervention indicated
  * G4: Life-threatening consequences; urgent intervention indicated
  * G5: Death
Wound infection | Up to 2 years after the completion of radiation therapy
  NIH-NCI Common Terminology Criteria for Adverse Events (CTCAE) Ver.5.0
  * G1: Localized, local intervention indicate
  * G2: Oral intervention indicated (e.g., antibiotic, antifungal, or antiviral)
  * G3: IV antibiotic, antifungal, or antiviral intervention indicated; invasive intervention indicated
  * G4: Life-threatening consequences; urgent intervention indicated
  * G5: Death
Wound Dehiscence | Up to 2 years after the completion of radiation therapy
  NIH-NCI Common Terminology Criteria for Adverse Events (CTCAE) Ver.5.0
  * G1: Incisional separation, intervention not indicated
  * G2: Incisional separation, local care (e.g., suturing) or medical intervention indicated (e.g., analgesic)
  * G3: Fascial disruption or dehiscence without evisceration; revision by operative intervention indicated
  * G4: Life-threatening consequences; symptomatic hernia with evidence of strangulation; fascial disruption with evisceration; major reconstruction flap, grafting, resection, or amputation indicated
  * G5: Death
Seroma | Up to 2 years after the completion of radiation therapy
  NIH-NCI Common Terminology Criteria for Adverse Events (CTCAE) Ver.5.0
  * G1: Asymptomatic; clinical or diagnostic observations only; intervention not indicated
  * G2: Symptomatic; simple aspiration indicated
  * G3: Symptomatic, elective invasive intervention indicated

OTHER OUTCOMES:
Arm Lymphedema [Optional] | Up to 2 years after the completion of radiation therapy
  In each follow-up time, arm circumference is measured at 10 cm above the ipsilateral and contralateral anterior cubital fossa. Lymphedema is considered to be occurred if a difference of ≥10% between two measures.
Cosmetic Outcome [Optional] | Up to 2 years after the completion of radiation therapy
  Skin 3D reconstruction was performed based on the radiation therapy plan CT and breast CT at 24 months after radiotherapy. Using in-house software based on deep learning algorithm, cosmetic scores are produced and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: In Ah Kim, MD. PhD., Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: No